CLINICAL TRIAL: NCT00702858
Title: Pilot, Single Center Randomized Controlled, Double-Blind, Cross Over, Intent to Treat Trial of Blue Citrus to Placebo in Those Breast Cancer Patients Receiving Aromatase Inhibitor Therapy
Brief Title: Trial of Blue Citrus Compared to Placebo in Patients Receiving Aromatase Inhibitor Therapy for Estrogen Receptor Positive Post-Menopausal Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Nathalie Johnson, Principal Investigator, Legacy Health System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Blue Citrus BC-AIT-001
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer; Joint Pain
Keywords: Breast Cancer; Joint Pain; Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms; Arthralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Blue Citrus either months 1-3 or 4-6
  Interventions: Drug: Blue Citrus
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Blue Citrus — Five 700 mg Capsules three times a day to equal 15 capsules per day for 3 months
  Arms: 1
Drug: Placebo — Five Placebo capsules three times a day to equal 15 capsules per day for 3 months
  Arms: 2

SUMMARY:
This purpose of this study is to determine if the herbal compound, Blue Citrus, decreases joint and bone pain associated with Aromotase Inhibitor therapy (AIT).

Another purpose of the study is to find out if Blue Citrus improves how you feel while taking AIT and if your quality of life improves.

DETAILED DESCRIPTION:
Post-menopausal women currently on AIT for breast cancer treatment who self-report musculoskeletal side effects related to AIT to their physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Post Menopausal - evidenced by no menses for the past 6 months or FSH level >40
2. Patient complaints of musculoskeletal symptoms
3. Currently taking AIT for ER positive postmenopausal breast cancer

Exclusion Criteria:

1. Previously taken Blue Citrus
2. Presence of bone metastasis
3. Unable to complete VAS Pain Scale
4. Unable to comply/complete SF 12 Quality of Life survey
5. Plan to discontinue AIT in less then six months
6. Unable to complete ADL scale
7. Have diagnosis of fibromyalgia
8. Have diagnosis of rheumatoid arthritis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine if Blue Citrus decreases musculoskeletal symptoms while on AIT as compared to Placebo | 6 months

SECONDARY OUTCOMES:
Determine if Blue Citrus use leads to reduction in use of other pain medications compared to placebo | 6 months
Determine if Blue Citrus compared to placebo improves Quality of Life,improves the ability to perform Activities of Daily Living | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Johnson, MD, Principal Investigator — Legacy Health System